CLINICAL TRIAL: NCT01299766
Title: Preventing Cognitive Decline in African Americans With Mild Cognitive Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Dartmouth College (Other); Johns Hopkins University (Other); University of Pennsylvania (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01AG035025 (NIH); 1R01AG035025 (NIH)
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Mild Cognitive Impairment; Memory
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavior Activation (Experimental): BA is a manual-based, behavioral treatment that helps people increase activity levels through goal setting, activity scheduling, graded task assignment, identifying avoidant behaviors, and rating one's sense of accomplishment.
  Interventions: Behavioral: Behavioral Activation (BA)
- Supportive Therapy (ST) (Placebo Comparator): ST is a person-centered treatment in which interventionists create a comfortable, non-judgmental environment by demonstrating genuineness, empathy, and acceptance of subjects without imposing any judgments on their decisions.
  Interventions: Behavioral: Supportive Therapy (ST)

INTERVENTIONS:
Behavioral: Behavioral Activation (BA) — BA is a manual-based, behavioral treatment that helps people increase activity levels through goal setting, activity scheduling, graded task assignment, identifying avoidant behaviors, and rating one's sense of accomplishment.
  Arms: Behavior Activation
Behavioral: Supportive Therapy (ST) — ST is a person-centered psychotherapy in which interventionists create a comfortable, non-judgmental environment by demonstrating genuineness, empathy, and acceptance of subjects without imposing any judgments on their decisions.
  Arms: Supportive Therapy (ST)

SUMMARY:
The goal of this study is to determine whether increasing participation in cognitive, physical, and/or social activities prevents cognitive decline in older African Americans (AAs) with Mild Cognitive Impairment (MCI). Patients with MCI are at increased risk for Alzheimer's Disease (AD); we propose that increasing participation in activities will prevent cognitive decline and may delay the onset of Alzheimer's Disease (AD). We will test this hypothesis by conducting a clinical trial in which older AAs with MCI (aged 65 years and older) will be randomized to Behavior Activation (BA) (a behavioral intervention that increases participation in daily activities) or Supportive Therapy (ST) (a person-centered psychotherapy that involves active listening and offering support focusing on participants' problems and concerns). We hypothesize that BA-treated subjects will have fewer declines in cognitive and functional abilities, fewer depressive and neuropsychiatric symptoms, and better quality of life than ST-treated subjects at 24 months.

DETAILED DESCRIPTION:
The goal of this study is to determine whether increasing participation in activities prevents cognitive decline in older African Americans with Mild Cognitive Impairment (MCI). We will attempt to increase activities with Behavioral Activation (BA). BA is a manual-based, behavioral treatment to increase activities as a way to improve function and mood. As patients do more (through activation) and perceive the benefit (i.e., feel better), their activity levels increase. BA promotes activities that reflect an individual's preferences and goals by structuring, scheduling, and reinforcing daily activities. This increases participation in activities with strong personal value, such as social engagement or normative role function, which in turn enhances mood and motivation to remain active.

The control treatment is Supportive Therapy, which is a non-directive, supportive therapy that is based on empathy, reflection, and support.

This study is specifically targeting older African Americans (AAs). Most clinical trials for MCI have tested pharmacologic treatments and have enrolled mostly Whites; their results may not apply to AAs whose life experiences and medical and genetic characteristics may exert unique effects. Those with MCI are a high-risk population for whom interventions to prevent cognitive decline are particularly important. Because AAs comprise one of the largest minority groups in the U.S., suffer disparities in health outcomes, and are unlikely to seek pharmacologic treatments or participate in clinical drug trials, there is an urgent need to enroll older AAs in non-pharmacologic intervention studies of cognition.

We will recruit 200 AA subjects aged 65 and older who have amnestic Mild Cognitive Impairment (MCI) - Multiple Domain subtype of MCI (aMCI-MD). One of the inclusion criteria is for participants to have a Knowledgeable Informant (KI) who is willing to participate in the study (with the subject's permission as documented in the informed consent form). A KI is defined as a family member or friend who is identified by the subject as someone who has regular and frequent contact with the subject (at least twice per week) in-person or by phone. The KI will be asked to provide information regarding the subject's functioning.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Having a friend/relative willing to serve as a Knowledgeable Informant (KI)
* Diagnosis of aMCI-MD
* Self-identified as African American

Exclusion Criteria:

* Psychiatric diagnosis, including dementia and major depression
* Sensory deficits that preclude neuropsychological testing
* Institutional residence
* Reduced life expectancy due to known terminal illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 221 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin J Casten, PhD, Study Director — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rovner BW, Casten RJ, Leiby B. Memory improvement in African Americans with amnestic mild cognitive impairment. Int J Geriatr Psychiatry. 2019 Oct;34(10):1447-1454. doi: 10.1002/gps.5141. Epub 2019 Jun 18. PMID 31087388
- [Derived] Rovner BW, Casten RJ, Hegel MT, Leiby B. Preventing Cognitive Decline in Black Individuals With Mild Cognitive Impairment: A Randomized Clinical Trial. JAMA Neurol. 2018 Dec 1;75(12):1487-1493. doi: 10.1001/jamaneurol.2018.2513. PMID 30208380
- [Derived] Rovner BW, Casten RJ. Preserving Cognition in Older African Americans with Mild Cognitive Impairment. J Am Geriatr Soc. 2016 Mar;64(3):659-61. doi: 10.1111/jgs.14012. No abstract available. PMID 27000348
- [Derived] Rovner BW, Casten RJ, Leiby BE. Determinants of Activity Levels in African Americans With Mild Cognitive Impairment. Alzheimer Dis Assoc Disord. 2016 Jan-Mar;30(1):41-6. doi: 10.1097/WAD.0000000000000096. PMID 25811797
- [Derived] Rovner BW, Casten RJ, Hegel MT, Leiby BE. Preventing cognitive decline in older African Americans with mild cognitive impairment: design and methods of a randomized clinical trial. Contemp Clin Trials. 2012 Jul;33(4):712-20. doi: 10.1016/j.cct.2012.02.016. Epub 2012 Mar 2. PMID 22406101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from June 21, 2011 to October 3, 2014; follow-up ended December 13, 2016. Potential participants were recruited when they sought memory screening at senior centers, senior housing sites, churches, and primary care clinics in Philadelphia, PA.
Pre-assignment Details: Prior to randomization, participants were administered neuropsychological tests to determine whether they met criteria for MCI. Participants with normal cognition and those with suspected dementia were excluded.
Period: Overall Study
Arm/Group | Behavior Activation | Supportive Therapy (ST)
Started | 111 | 110
Completed (Provided data at 24 months) | 77 | 87
Not Completed | 34 | 23
Not completed — Death | 5 | 4
Not completed — Withdrawal by Subject | 29 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavior Activation | Supportive Therapy (ST) | Total
Number analyzed (Participants) | 111 | 110 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.5 (7.1) | 76.2 (6.9) | 75.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 89 | 175
  Male | 25 | 21 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 110 | 110 | 220
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 111 | 110 | 221
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 111 | 110 | 221

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decline of 6 Points on the Hopkins Verbal Learning Test-Revised (HVLT-R)
Description: A decline of 6 points from baseline to 24 months on the Hopkins Verbal Learning Test-Revised (HVLT-R). Possible scores range from 0 to 12, with higher scores indicating better memory.
Time Frame: 24 months
Population: The primary analysis was performed on the modified intent to treat population including all available data from all participants with at least one follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavior Activation | Supportive Therapy (ST)
Number analyzed (Participants) | 91 | 99
Participants | 1 | 9
Statistical Analysis 1: Comparison: Behavior Activation vs Supportive Therapy (ST); Poisson regression with robust standard errors (GEE) was used to jointly model decline in HVLT-R Total Recall score ≥ 6 words at 6, 12, 18, and 24 months by treatment group. The model included time, treatment, time-by-treatment interaction terms, and baseline HVLT-R Total Recall score; Test type: Superiority; p = .02, Poisson regression with robust SE (GEE); Risk Ratio (RR) = 0.12, 95% CI 2-sided [0.02 to 0.74]

2. Secondary Outcome: Change in University of California Performance-based Skills Assessment (UPSA) Score Per Year
Description: The University of California Performance-based Skills Assessment (UPSA) was used as an objective test of accuracy with writing checks, making change, using a telephone, and scheduling a physician appointment (higher scores indicate better function). Possible scores range from 0 to 100.
Time Frame: 24 months
Population: The analysis was performed on the modified intent to treat population including all available data from all participants with at least one follow-up visit.
Measure: Mean (95% Confidence Interval); unit: units per year
Arm/Group | Behavior Activation | Supportive Therapy (ST)
Number analyzed (Participants) | 91 | 99
units per year | -.13 [-2.05 to 1.79] | -2.60 [-4.36 to -0.83]
Statistical Analysis 1: Comparison: Behavior Activation vs Supportive Therapy (ST); Mixed effects linear regression was used to model the trajectory. Fixed effects for time (as a continuous variable), treatment group, time-by-treatment group interaction, and age at baseline were included. Random intercepts and slopes were included to account for within-subject correlation; Test type: Superiority; p = .064, Mixed Models Analysis; Difference in Slopes = 2.47, 95% CI 2-sided [-.14 to 5.07]

ADVERSE EVENTS:
Time Frame: 2 years
Description: We reported hospitalizations
Arm/Group | Behavior Activation | Supportive Therapy (ST)
All-Cause Mortality (participants affected / at risk) | 5/111 | 4/110
Serious Adverse Events (participants affected / at risk) | 40/111 | 35/110
Other Adverse Events (participants affected / at risk) | 0/111 | 0/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavior Activation (N=111) | Supportive Therapy (ST) (N=110)
Death (Infections and infestations) | 0 (0) | 1 (1) — Death from septic shock
Death NOS (Investigations) | 5 (5) | 4 (4) — Death NOS
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fractured disk
Broken shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chrohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hernia repair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Valve replacement (Cardiac disorders) | 1 (1) | 1 (1)
Pacemaker implanted (Cardiac disorders) | 2 (2) | 1 (1)
Seziure (Nervous system disorders) | 1 (1) | 0 (0)
UTI (Infections and infestations) | 0 (0) | 3 (3)
Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Heart attack (Cardiac disorders) | 2 (2) | 1 (1)
Stroke (Vascular disorders) | 4 (4) | 4 (5)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Renal and urinary disorders) | 0 (0) | 2 (2)
bypass surgery (Cardiac disorders) | 2 (2) | 0 (0)
hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blood clot (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
CHF (Cardiac disorders) | 1 (1) | 0 (0)
GI symptoms (Gastrointestinal disorders) | 2 (2) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Knee replacement (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
internal bleeding (Eye disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The racial characteristics of the sample and motivation to enroll a clinical trial, limit generalizability. Also, nonrandom attrition (higher in males) may have skewed results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No